CLINICAL TRIAL: NCT01605474
Title: Safety, Efficacy, and Patient Satisfaction of Cervical Ripening With Transcervical Use of the Foley Catheter in an Outpatient Setting
Brief Title: Patient Satisfaction of Cervical Ripening in an Outpatient Setting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Gregory W. Lau, MD, Fellow, Maternal Fetal Medicine, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00026352
Record Dates: First submitted 2012-05-18; First posted 2012-05-25 (Estimated); Last update posted 2012-05-25 (Estimated); Status verified 2012-05

CONDITIONS: Pregnancy
Keywords: foley catheter; foley bulb; induction of labor; labor
MeSH Terms: interventions — Inosine Monophosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Outpatient Cervical Ripening (Active Comparator): Patients who are randomized to this arm will be allowed discharged home for 12 hours after fetal status is assessed and noted to be reassuring with the foley bulb in place. They will return sooner if they experience rupture of membranes or enter active labor or if the foley bulb falls out.
  Interventions: Other: Patient discharged home after foley bulb placement.
- Inpatient Cervical Ripening (No Intervention): In this arm, the fetus will be assessed and a foley bulb placed but these patients will be kept in the hospital.
  Interventions: Other: Inpatient

INTERVENTIONS:
Other: Patient discharged home after foley bulb placement. — The patient will be discharged home after fetal status is evaluated and noted to be reassuring. A 16 French foley bulb insufflated with 30 cc of normal saline will be placed and secured to the patient's inner thigh.
  Other Names: Foley bulb (16 French)
  Arms: Outpatient Cervical Ripening
Other: Inpatient — The patients will not be discharged home after assessment and placement of the foley catheter.
  Other Names: Foley Bulb (16 French)
  Arms: Inpatient Cervical Ripening

SUMMARY:
This study examines whether outpatient pre-induction cervical ripening improves patient satisfaction and is safe and effective.

DETAILED DESCRIPTION:
Objective:

To compare inpatient versus outpatient preinduction cervical ripening in order to evaluate differences between each setting with respect to patient safety, satisfaction and cesarean rate.

Background:

Many women who require induction of labor present with an unripe cervix. This has been associated with a longer duration of labor as well as higher rates of failed induction resulting in cesarean delivery. These patients are also at higher risk for postpartum hemorrhage, blood transfusion, and cesarean hysterectomy. Preinduction cervical ripening is thought to improve the likelihood of a successful induction in women with an unripe cervix. Prolonged inductions of labor do not only lead to patient dissatisfaction but also use valuable resources such as available labor and delivery bed and nursing staff. This in turn overburdens labor and delivery resources which are already taxed. These issues contribute to increasing costs as well as decreasing patient satisfaction.

Prior studies have shown that moving preinduction cervical ripening from an inpatient setting to an outpatient setting can decrease costs significantly. It is also thought that 50% of all patients requiring induction of labor may be eligible for outpatient cervical ripening. Many of these studies have looked at PGE two preparations which are no longer commonly used. However, a study by Scisione et al. from November 2001 looked at the use of Trent cervical Foley catheter for this purpose. They had previously shown that a mechanical method, the Foley catheter, had significant advantages over preparations such as prepidil. Scisione et al. had also previously shown that in a randomized trial comparing misoprostol and Foley catheter for preinduction cervical ripening both were found to be equally effective. However, in the group who received the misoprostol, there was an increased risk of meconium passage in uterine contractile abnormalities.

The Foley catheter appears to be safe and efficacious. It also appears to be a good option for outpatient preinduction cervical ripening. One of the downsides of using a Foley catheter for preinduction cervical ripening is that it requires checking and readjusting. The economic benefits of outpatient cervical ripening and the social advantages for patients seem very promising. However, many women may need to return to the hospital as a result of anxiety or questions surrounding the use of the Foley catheter for preinduction cervical ripening.

In the study by Scisione et al. which involved 111 women, the primary outcome variable was a change in Bishop score. There was no statistically significant difference noted with respect to each of the groups. There were also no statistically significant differences with respect to a maximum dose of oxytocin used subsequently in labor nor was there a difference in the amount of time the Pitocin was used. No statistically significant differences were noted in the total induction times, cesarean delivery rates, and NICU admissions, Apgar scores or birth weights between groups. There were differences noted in the preinduction cervical ripening times between the different groups. Notably, the outpatient group had a longer preinduction cervical ripening time.

In the aforementioned study, patients were asked to describe their discomfort during the preinduction cervical ripening phase using a visual analog test. This is based on a scale of 1 to 10 where 1 was noted as no discomfort or minimal discomfort and 10 was the worst pain imaginable. The outpatient group reported a median discomfort level of 4.8 where the inpatient group reported a discomfort level 3.9. These results were not statistically significant. Most of the discomfort was noted during Foley catheter placement.

With respect to the cesarean delivery rates between groups it is of note that there is a decrease noted by the authors of the study in the patients who underwent the outpatient cervical ripening versus those who underwent the inpatient cervical ripening. The authors of the study are unclear of the reason for this difference. However, this study was underpowered to detect this difference given that 284 patients would be needed in each group to reach adequate power to state whether the differences noted between groups is significant.

Demographically, there were no statistically significant differences between groups with respect maternal age, gravidity, distasteful age, amniotic fluid index, source of insurance. Based on the results of this study, if both methods are equally efficacious but the outpatient method leads to higher patient satisfaction, decreases inpatient resource use and leads to a decreased cesarean rate, it may be the preferred method of preinduction cervical ripening. Based on this hypothesis, the investigators would like to compare the use of the foley catheter for preinduction cervical ripening in an inpatient versus outpatient setting with respect to patient safety, satisfaction and cesarean rate.

At Cedars-Sinai, there are approximately 7000 deliveries per year. The induction rate approximates 22% which results in 1540 inductions per year. At the present time, these are all inpatients. Outpatient cervical ripening is not standard of care at Cedars-Sinai but it has been evaluated at other institutions and its safety has been validated. Advantages of an outpatient pre-induction cervical ripening includes shorter hospital stays, decreased cesarean section rates, improved patient comfort and satisfaction. With a reduced cesarean section rate, there is also the potential for decreased NICU admissions.

With respect to potential risks of an outpatient induction, they are similar to that of inpatient inductions. Risks of this procedure include rupture of amniotic membranes and active labor. Both of which would result in admission and delivery.

Methods:

A randomized controlled trial is planned in women with a term gestation in the vertex presentation, a reactive nonstress test, an amniotic fluid index above five, and a Bishop score of no more than five. The primary outcome variable will be a change in Bishop score as well as patient satisfaction. The secondary outcome will be change in cesarean section rates. There will be two groups in the study: those who undergo inpatient cervical ripening and those who undergo outpatient cervical ripening. A Foley catheter with a 30 mL balloon will be placed through the cervix on gentle traction in each group in the usual fashion that is currently used.

The outpatient group will be discharged home with written instructions. These patients will also be instructed to return 12 hours after placement for their induction. The inpatient group will be kept in the hospital during the same time period for their cervical ripening.

Exclusion criteria include the following: placenta previa and/or accreta, low lying placenta, undiagnosed vaginal bleeding, preeclampsia, fetal anomaly, intrauterine growth restriction, RH isoimmunization, fetal demise, rupture of membranes, maternal heart disease, known latex allergy, active genital herpes infection, previous uterine surgery, limited access to a telephone, excessive distance from the hospital, and/ or unreliable transportation.

Upon presentation to labor and delivery an initial assessment will be conducted and the history and physical examination completed by the house staff. An amniotic fluid index would also be obtained and if the amniotic fluid index is less than five the patient would not be considered a candidate for the study. If the patient remains a candidate, the procedure for Foley catheter placement will be explained to the patient. Prior to placement of the Foley, a digital exam will be performed and a Bishop score assigned by the attending or senior-level resident. A number 16 Foley catheter with a 30 mL balloon will be inserted into the endocervical canal under direct visualization via a speculum exam or by blind placement. The Foley catheter will be advanced to or passed through the internal os and subsequently filled with 30 mL of sterile water. The catheter will then be placed on gentle traction by taping the catheter to the medial portion of the thigh. The nonstress test will be performed before and after Foley catheter placement. If the fetal heart rate is reactive and there is no sign of uterine tachysystole, uterine hypertonus or non-reassuring fetal testing, then the patient will be randomized to either group.

ELIGIBILITY:
Inclusion Criteria:

* term pregnancy
* singleton gestation
* cephalic presentation
* scheduled for an induction of labor (acceptable conditions include gestational diabetes, chronic hypertension)

Exclusion criteria include the following:

* placenta previa and/or accreta
* low lying placenta
* undiagnosed vaginal bleeding
* preeclampsia
* fetal anomaly
* intrauterine growth restriction
* RH isoimmunization
* fetal demise
* rupture of membranes
* maternal heart disease
* known latex allergy
* active genital herpes infection
* previous uterine surgery
* limited access to a telephone
* excessive distance from the hospital, and/or
* unreliable transportation

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 800 (Estimated)
Dates: Start 2012-04; Primary Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Cesarean section rate | 2 years
  Cesarean delivery rate between groups

SECONDARY OUTCOMES:
Patient satisfaction (Pain /discomfort) | 2 year
  Patient satisfaction. Administering a questionaire on which the patient will rate her pain/discomofrt during the placement of the foley bulb and her pain/discomfort while undergoing labor. The Wong Baker Faces scale will be used to assess this measure.
Apgar scores | 2 years
  Apgar scores
NICU admissions | 2 years
  Neonatal ICU admissions after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Tania Esaoff, MD, Principal Investigator — Cedars-Sinai Medical Center, Department of Obstetrics and Gynecology, Division of Maternal Fetal Medicine
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Background] Sciscione AC, Muench M, Pollock M, Jenkins TM, Tildon-Burton J, Colmorgen GH. Transcervical Foley catheter for preinduction cervical ripening in an outpatient versus inpatient setting. Obstet Gynecol. 2001 Nov;98(5 Pt 1):751-6. doi: 10.1016/s0029-7844(01)01579-4. PMID 11704164